CLINICAL TRIAL: NCT01968772
Title: Effect of Transdermal Magnesium Chloride on Quality of Life in Patients With Fibromyalgia - A Pilot Study
Brief Title: Effect of Transdermal Magnesium Chloride on Quality of Life in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Magnesium Direct (Unknown)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-001413
Record Dates: First submitted 2013-04-04; First posted 2013-10-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia; Fibromyalgia Syndrome
Keywords: Fibromyalgia; Fibromyalgia Syndrome; Magnesium Chloride; Transdermal Magnesium Chloride
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transdermal Magnesium Chloride (Other): This is a clear, odorless liquid that dries rapidly on the skin and leaves no oily residue. Its ingredients are water, magnesium chloride, and a proprietary blend of less than two-tenths of 1% trace minerals (Boron, Selenium, and Manganese).
  Interventions: Other: Transdermal Magnesium Chloride

INTERVENTIONS:
Other: Transdermal Magnesium Chloride — Each participant will be provided with a spray bottle containing a transdermal magnesium chloride solution and asked to apply 4 sprays per each arm and each leg 2 times a day as follows: pump 4 sprays into the palm of your hand and apply to each arm and each leg 2 times a day for a total of 32 sprays daily. Rub the contents of 4 sprays on one limb and repeat for each limb coating evenly.

SUMMARY:
In this pilot study we propose to gather preliminary data on whether transdermal magnesium chloride can improve quality of life in patients with fibromyalgia. Forty women with fibromyalgia will be enrolled in this study. Participants will be asked to apply a topical solution of magnesium chloride on their extremities 3 times daily for 28 consecutive days. Three questionnaires measuring quality of life will be administered at baseline, at 2 weeks, and at 4 weeks (end of study).

DETAILED DESCRIPTION:
Fibromyalgia is a chronic pain syndrome with no known etiology. Fibromyalgia is generally diagnosed in patients reporting widespread musculoskeletal pain, and tenderness. In addition to widespread pain, fibromyalgia is also characterized by chronic fatigue, depression, sleep disturbances, and poor concentration. It has been reported that approximately 3.5% of women and 0.5% of men in the United States suffer from fibromyalgia. While the primary cause of fibromyalgia remains unclear, a growing body of evidence indicates that the widespread pain associated with fibromyalgia is due to abnormalities in the central nervous system. The pain threshold, both mechanical and thermal, in fibromyalgia sufferers are lowered such that it requires a lesser than normal stimulus to elicit pain.

Recent reports suggest that fibromyalgia is an oxidative stress disorder and deficiency in trace elements and antioxidants play an important role in the development of fibromyalgia. Magnesium is a trace element that is important for many metabolic functions. It affects cell membrane permeability and electrical activity. The similarity in the clinical symptoms of fibromyalgia and magnesium deficiency along with the histopathological findings of tender points (such as hypoxia and adenosine triphosphate deficiency) raises the possibility that magnesium may play a role in fibromyalgia etiopathogenesis.

In this pilot study we propose to explore the feasibility and ease of 2 times a day application of a topical solution to the arms and legs. We will also gather preliminary data on whether transdermal magnesium chloride can improve quality of life in women with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with fibromyalgia at Mayo Clinic Rochester's Fibromyalgia Clinic
* Postmenopausal women (no menstrual period for 1 year or more)
* Women age 40-70 that have had a hysterectomy
* Willing to travel to Mayo Clinic Rochester for the initial instruction visit
* Able to apply the transdermal magnesium chloride as directed
* Able to complete the questionnaires and daily diary
* Able and willing to give informed consent
* Able to speak, write and understand English

Exclusion Criteria:

* Patients on dialysis
* Individuals who decline to participate in the study
* Diagnoses of bipolar disorder, schizophrenia or dementia
* Patients with myasthenia gravis and myasthenic syndromes
* Patients on magnesium supplements

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of study on quality of life as documented by the Revised Fibromyalgia Impact Questionnaire (FIQR) in women with fibromyalgia after applying a transdermal magnesium chloride solution to their arms and legs 2 times daily. | 28 Days

SECONDARY OUTCOMES:
Change from baseline to study end on quality of life as documented by the SF-36v2 Health Survey in women with fibromyalgia after applying a transdermal magnesium chloride solution to their extremities 2 times daily. | 28 Days
Change from baseline to study end on quality of life as documented by the Quality of Life Analog Scale (QOL Analog Scale) in women with fibromyalgia after applying a transdermal magnesium chloride solution to their extremities 2 times daily. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Dietlind L. Wahner-Roedler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Goldenberg DL, Burckhardt C, Crofford L. Management of fibromyalgia syndrome. JAMA. 2004 Nov 17;292(19):2388-95. doi: 10.1001/jama.292.19.2388. PMID 15547167
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Wolfe F, Cathey MA. Prevalence of primary and secondary fibrositis. J Rheumatol. 1983 Dec;10(6):965-8. PMID 6582268
- [Background] Wolfe F, Cathey MA. The epidemiology of tender points: a prospective study of 1520 patients. J Rheumatol. 1985 Dec;12(6):1164-8. PMID 3879278
- [Background] Staud R, Vierck CJ, Cannon RL, Mauderli AP, Price DD. Abnormal sensitization and temporal summation of second pain (wind-up) in patients with fibromyalgia syndrome. Pain. 2001 Mar;91(1-2):165-75. doi: 10.1016/s0304-3959(00)00432-2. PMID 11240089
- [Background] Banic B, Petersen-Felix S, Andersen OK, Radanov BP, Villiger PM, Arendt-Nielsen L, Curatolo M. Evidence for spinal cord hypersensitivity in chronic pain after whiplash injury and in fibromyalgia. Pain. 2004 Jan;107(1-2):7-15. doi: 10.1016/j.pain.2003.05.001. PMID 14715383
- [Background] Ali M, Ali O. Fibromyalgia: An oxidative-dysoxygenative disorder (ODD). J Integr Med. 1999;3:17-37.
- [Background] Bagis S, Tamer L, Sahin G, Bilgin R, Guler H, Ercan B, Erdogan C. Free radicals and antioxidants in primary fibromyalgia: an oxidative stress disorder? Rheumatol Int. 2005 Apr;25(3):188-90. doi: 10.1007/s00296-003-0427-8. Epub 2003 Dec 20. PMID 14689230
- [Background] Chung CP, Titova D, Oeser A, Randels M, Avalos I, Milne GL, Morrow JD, Stein CM. Oxidative stress in fibromyalgia and its relationship to symptoms. Clin Rheumatol. 2009 Apr;28(4):435-8. doi: 10.1007/s10067-008-1072-0. Epub 2008 Dec 17. PMID 19089486
- [Background] Iqbal R, Mughal MS, Arshad N, Arshad M. Pathophysiology and antioxidant status of patients with fibromyalgia. Rheumatol Int. 2011 Feb;31(2):149-52. doi: 10.1007/s00296-010-1470-x. Epub 2010 Apr 8. PMID 20376669
- [Background] London M. The role of magnesium in fibromyalgia. 1994. http://web.mit.edu/london/www.magnesium.html
- [Background] Magaldi M, Moltoni L, Biasi G, Marcolongo R. [Changes in intracellular calcium and magnesium ions in the physiopathology of the fybromyalgia syndrome]. Minerva Med. 2000 Jul-Aug;91(7-8):137-40. Italian. PMID 11155461
- [Background] Eisinger J, Zakarian H, Pouly E, Plantamura A, Ayavou T. Protein peroxidation, magnesium deficiency and fibromyalgia. Magnes Res. 1996 Dec;9(4):313-6. PMID 9247880
- [Background] Clauw D, Ward K, Katz P, Rajan S. Muscle intracellular magnesium levels with pain tolerance in fibromyalgia (FM). Arthritis Rheumat. 1994;S213:324.
- [Derived] Engen DJ, McAllister SJ, Whipple MO, Cha SS, Dion LJ, Vincent A, Bauer BA, Wahner-Roedler DL. Effects of transdermal magnesium chloride on quality of life for patients with fibromyalgia: a feasibility study. J Integr Med. 2015 Sep;13(5):306-13. doi: 10.1016/S2095-4964(15)60195-9. PMID 26343101